CLINICAL TRIAL: NCT03510234
Title: Self-confidence Study in Patients With Argus II Artificial Retina
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6954
Record Dates: First submitted 2018-02-26; First posted 2018-04-27 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-02

CONDITIONS: Pigmentary Retinopathy
Keywords: Pigmentary retinopathy; Argus II retinal prosthesis; Self-confidence
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate whether the use of the Argus II retinal prosthesis improves the confidence and self-esteem of patients with advanced retinopathy pigmentosa

ELIGIBILITY:
Inclusion Criteria:

* Major patient (≥18 years old)
* Patient already operated in France with artificial retina and having 1 year of follow-up
* Patient who has agreed to use his medical data for research purposes

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient already operated in France with artificial retina and having 1 year of follow-up
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Self-confidence | 12 months
  Evaluation of Self-confidence via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David GAUCHER, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service D'Ophtalmologie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No